CLINICAL TRIAL: NCT01358864
Title: A Phase III, Randomised, Double-blind and Placebo Controlled Study of Once Daily BI 201335, 240 mg for 12 or 24 Weeks in Combination With Pegylated interferon-a (PegIFNa) and Ribavirin (RBV) in Patients With Genotype 1 Chronic Hepatitis C Infection Who Failed a Prior PegIFN/RBV Treatment
Brief Title: Efficacy and Safety of BI 201335 (Faldaprevir) in Combination With Pegylated Interferon-alpha and Ribavirin in Treatment-Experienced Genotype 1 Hepatitis C Infected Patients (STARTverso 3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1220.7; 2010-021715-17 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-05-23; First posted 2011-05-24 (Estimated); Results first posted 2015-10-28 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — faldaprevir; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo/PegIFN/RBV (Active Comparator): patient to receive two capsules identical to those containing BI201335 once a day for 24 weeks and PegIFN/RBV for 48 weeks
  Interventions: Drug: Pegylated Interferon-alpha (IFN); Drug: Ribavirin (RBV); Drug: Placebo
- BI201335 12 weeks (Experimental): patient to receive two capsules containing BI 201335 once a day for 12 weeks and PegIFN/RBV for 48 weeks
  Interventions: Drug: BI 201335; Drug: Pegylated Interferon-alpha (IFN); Drug: Ribavirin (RBV)
- BI201335 24 weeks (Experimental): patient to receive two capsules containing BI 201335 once a day for 24 weeks and PegIFN/RBV for 48 weeks
  Interventions: Drug: BI 201335; Drug: Pegylated Interferon-alpha (IFN); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: BI 201335 — BI 201335 once a day (QD) for 24 weeks
  Arms: BI201335 12 weeks; BI201335 24 weeks
Drug: Pegylated Interferon-alpha (IFN) — Pegylated Interferon-alpha for 48 weeks
Drug: Ribavirin (RBV) — Ribavirin (RBV) for 24 or 48 weeks
Drug: Placebo — Placebo to BI201335 for 24 weeks
  Arms: Placebo/PegIFN/RBV

SUMMARY:
The aim of this trial is to evaluate the efficacy and the safety of BI 201335 given for 12 or 24 weeks in combination with PegIFN/RBV given for 48 weeks as compared to PegIFN/RBV alone in chronic GT-1 hepatitis C virus infected patients who failed a prior PegIFN/RBV treatment.

ELIGIBILITY:
Inclusion criteria:

1. Chronic hepatitis C genotype 1 infection, diagnosed at least 6 months prior to screening
2. Confirmed prior virological failure with an approved dose of PegIFN/RBV
3. Age 18 to 70 years,
4. HCV RNA (RiboNucleic Acid) = 1,000 IU/mL at screening,

Exclusion criteria:

1. HCV infection of mixed genotype; Hepatitis B Virus (HBV) or Human Immunodeficiency Virus (HIV) co-infection
2. Evidence of acute or chronic liver disease due to causes other than chronic HCV infection,
3. Decompensated liver disease, or history of decompensated liver disease,
4. Body weight < 40 or > 125 kg,
5. Clinical evidence of significant or unstable cardiovascular disease, chronic pulmonary disease, history or evidence of retinopathy or clinically significant ophthalmological disorder
6. Pre-existing psychiatric condition that could interfere with the subject's participation in and completion of the study
7. Laboratory parameters disorders (thalassemia major, sickle cell anemia or G6PD deficit)
8. Hemoglobin < 12 g/dL for women and < 13 g/dL for men
9. Patients who have been previously treated with at least one dose of any antiviral or immunomodulatory drug other than interferon alfa or ribavirin for acute or chronic HCV infection including and not restricted to protease or polymerase inhibitors,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 678 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (116):
- United States (18):
  - 1220.7.0091 Boehringer Ingelheim Investigational Site, North Little Rock, Arkansas
  - 1220.7.0082 Boehringer Ingelheim Investigational Site, Englewood, Colorado
  - 1220.7.0095 Boehringer Ingelheim Investigational Site, Palm Harbor, Florida
  - 1220.7.0039 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 1220.7.0013 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1220.7.0062 Boehringer Ingelheim Investigational Site, Vaiparaiso, Indiana
  - 1220.7.0085 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 1220.7.0087 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 1220.7.0101 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1220.7.0027 Boehringer Ingelheim Investigational Site, Framingham, Massachusetts
  - 1220.7.0012 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.7.0077 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1220.7.0058 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1220.7.0063 Boehringer Ingelheim Investigational Site, Arlington, Texas
  - 1220.7.0029 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1220.7.0071 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1220.7.0009 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1220.7.0016 Boehringer Ingelheim Investigational Site, San Antonio, Texas
- Austria (3):
  - 1220.7.4303 Boehringer Ingelheim Investigational Site, Linz
  - 1220.7.4301 Boehringer Ingelheim Investigational Site, Vienna
  - 1220.7.4302 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (7):
  - 1220.7.3201 Boehringer Ingelheim Investigational Site, Brussels
  - 1220.7.3207 Boehringer Ingelheim Investigational Site, Brussels
  - 1220.7.3204 Boehringer Ingelheim Investigational Site, Edegem
  - 1220.7.3205 Boehringer Ingelheim Investigational Site, Ghent
  - 1220.7.3206 Boehringer Ingelheim Investigational Site, Jette
  - 1220.7.3202 Boehringer Ingelheim Investigational Site, Leuven
  - 1220.7.3203 Boehringer Ingelheim Investigational Site, Liège
- Canada (9):
  - 1220.7.1011 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 1220.7.1012 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1220.7.1003 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1220.7.1016 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1220.7.1007 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1220.7.1004 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1220.7.1006 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1220.7.1010 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 1220.7.1014 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- France (12):
  - 1220.7.3301 Boehringer Ingelheim Investigational Site, Clichy
  - 1220.7.3311 Boehringer Ingelheim Investigational Site, Lille
  - 1220.7.3303 Boehringer Ingelheim Investigational Site, Marseille
  - 1220.7.3304 Boehringer Ingelheim Investigational Site, Montpellier
  - 1220.7.3305 Boehringer Ingelheim Investigational Site, Nice
  - 1220.7.3302 Boehringer Ingelheim Investigational Site, Paris
  - 1220.7.3310 Boehringer Ingelheim Investigational Site, Paris
  - 1220.7.3316 Boehringer Ingelheim Investigational Site, Pessac
  - 1220.7.3317 Boehringer Ingelheim Investigational Site, Reims
  - 1220.7.3315 Boehringer Ingelheim Investigational Site, Rennes
  - 1220.7.3318 Boehringer Ingelheim Investigational Site, Strasbourg
  - 1220.7.3308 Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy
- Germany (11):
  - 1220.7.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.7.4904 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.7.4913 Boehringer Ingelheim Investigational Site, Dortmund
  - 1220.7.4906 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1220.7.4901 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1220.7.4908 Boehringer Ingelheim Investigational Site, Hamburg
  - 1220.7.4918 Boehringer Ingelheim Investigational Site, Hanover
  - 1220.7.4907 Boehringer Ingelheim Investigational Site, Herne
  - 1220.7.4903 Boehringer Ingelheim Investigational Site, Leipzig
  - 1220.7.4911 Boehringer Ingelheim Investigational Site, Mainz
  - 1220.7.4905 Boehringer Ingelheim Investigational Site, München
- Japan (24):
  - 1220.7.8106 Boehringer Ingelheim Investigational Site, Chiba, Chiba
  - 1220.7.8111 Boehringer Ingelheim Investigational Site, Gifu, Gifu
  - 1220.7.8107 Boehringer Ingelheim Investigational Site, Itabashi-ku, Tokyo
  - 1220.7.8112 Boehringer Ingelheim Investigational Site, Izunokuni, Shizuoka
  - 1220.7.8108 Boehringer Ingelheim Investigational Site, Kamakura, Kanagawa
  - 1220.7.8117 Boehringer Ingelheim Investigational Site, Kita-gun, Kagawa
  - 1220.7.8109 Boehringer Ingelheim Investigational Site, Kofu, Yamanashi
  - 1220.7.8116 Boehringer Ingelheim Investigational Site, Kurashiki, Okayama
  - 1220.7.8118 Boehringer Ingelheim Investigational Site, Kurume, Fukuoka
  - 1220.7.8110 Boehringer Ingelheim Investigational Site, Matsumoto, Nagano
  - 1220.7.8124 Boehringer Ingelheim Investigational Site, Matsuyama, Ehime
  - 1220.7.8113 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1220.7.8105 Boehringer Ingelheim Investigational Site, Namegata, Ibaraki
  - 1220.7.8114 Boehringer Ingelheim Investigational Site, Nishinomiya, Hyogo
  - 1220.7.8125 Boehringer Ingelheim Investigational Site, Ogaki, Gifu
  - 1220.7.8119 Boehringer Ingelheim Investigational Site, Omura, Nagasaki
  - 1220.7.8122 Boehringer Ingelheim Investigational Site, Omuta, Fukuoka
  - 1220.7.8121 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1220.7.8101 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1220.7.8102 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1220.7.8115 Boehringer Ingelheim Investigational Site, Tanabe, Wakayama
  - 1220.7.8123 Boehringer Ingelheim Investigational Site, Toyama,Toyama
  - 1220.7.8126 Boehringer Ingelheim Investigational Site, Tsu, Mie
  - 1220.7.8104 Boehringer Ingelheim Investigational Site, Tsuchiura, Ibaraki
- Portugal (6):
  - 1220.7.3503 Boehringer Ingelheim Investigational Site, Aveiro
  - 1220.7.3509 Boehringer Ingelheim Investigational Site, Barreiro
  - 1220.7.3506 Boehringer Ingelheim Investigational Site, Coimbra
  - 1220.7.3501 Boehringer Ingelheim Investigational Site, Lisbon
  - 1220.7.3505 Boehringer Ingelheim Investigational Site, Lisbon
  - 1220.7.3502 Boehringer Ingelheim Investigational Site, Porto
- 1220.7.0034 Boehringer Ingelheim Investigational Site, San Juan, Puerto Rico
- Spain (12):
  - 1220.7.3406 Boehringer Ingelheim Investigational Site, A Coruña
  - 1220.7.3402 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.7.3404 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.7.3411 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.7.3412 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.7.3405 Boehringer Ingelheim Investigational Site, Madrid
  - 1220.7.3409 Boehringer Ingelheim Investigational Site, Madrid
  - 1220.7.3410 Boehringer Ingelheim Investigational Site, Majadahonda-Madrid
  - 1220.7.3408 Boehringer Ingelheim Investigational Site, Santander
  - 1220.7.3403 Boehringer Ingelheim Investigational Site, Seville
  - 1220.7.3401 Boehringer Ingelheim Investigational Site, Valencia
  - 1220.7.3407 Boehringer Ingelheim Investigational Site, Vigo (Pontevedra)
- Switzerland (5):
  - 1220.7.4106 Boehringer Ingelheim Investigational Site, Bern
  - 1220.7.4103 Boehringer Ingelheim Investigational Site, La Chaux-de-Fonds
  - 1220.7.4107 Boehringer Ingelheim Investigational Site, Lugano
  - 1220.7.4108 Boehringer Ingelheim Investigational Site, Sankt Gallen
  - 1220.7.4101 Boehringer Ingelheim Investigational Site, Zurich
- United Kingdom (8):
  - 1220.7.4405 Boehringer Ingelheim Investigational Site, Bristol
  - 1220.7.4404 Boehringer Ingelheim Investigational Site, London
  - 1220.7.4409 Boehringer Ingelheim Investigational Site, London
  - 1220.7.4410 Boehringer Ingelheim Investigational Site, London
  - 1220.7.4401 Boehringer Ingelheim Investigational Site, Manchester
  - 1220.7.4408 Boehringer Ingelheim Investigational Site, Nottingham
  - 1220.7.4407 Boehringer Ingelheim Investigational Site, Oxford
  - 1220.7.4403 Boehringer Ingelheim Investigational Site, Southampton

RESULTS

PARTICIPANT FLOW:
Groups:
- Relapser:Placebo: Patients who had had a prior relapse, received 2 soft gelatin capsules identical to those containing Faldaprevir once daily (orally) and PegIFN/RBV (Pegylated interferon alpha-2a/Ribavirin) administered by injection, for 24 weeks, followed by PegIFN/RBV for 24 weeks.
- Relapser:Faldaprevir 12 Weeks: Patients who had had a prior relapse, received Faldaprevir (BI 201335) 240mg once daily, in the form of 2 soft gelatin capsules administered orally, combined with PegIFN/RBV, administered by injection, for 12 weeks, followed by placebo once daily combined with PegIFN/RBV for 12 weeks. At week 24, if the patients did not achieve early treatment success (ETS) the patients received an additional 24 weeks of PegIFN/RBV alone.
- Relapser:Faldaprevir 24 Weeks: Patients who had had a prior relapse, received Faldaprevir 240mg once daily, in the form of 2 soft gelatin capsules administered orally, combined with PegIFN/RBV, administered by injection, for 24 weeks. At week 24, if the patients did not achieve early treatment success (ETS) the patients received an additional 24 weeks of PegIFN/RBV alone.
- Partial:Placebo: Patients who had had a prior partial response, received 2 soft gelatin capsules identical to those containing Faldaprevir once daily (orally) and PegIFN/RBV (Pegylated interferon alpha-2a/Ribavirin) administered by injection, for 24 weeks, followed by PegIFN/RBV for 24 weeks.
- Partial:Faldaprevir 12 Weeks: Patients who had had a prior partial response, received Faldaprevir 240mg once daily, in the form of 2 soft gelatin capsules administered orally, combined with PegIFN/RBV, administered by injection, for 12 weeks, followed by placebo once daily combined with PegIFN/RBV for 12 weeks. Followed by PegIFN/RBV alone for 24 weeks.
- Partial:Faldaprevir 24 Weeks: Patients who had had a prior partial response, received Faldaprevir 240mg once daily, in the form of 2 soft gelatin capsules administered orally, combined with PegIFN/RBV, administered by injection, for 24 weeks. Followed by PegIFN/RBV alone for 24 weeks.
- Null:Faldaprevir 12 Weeks: Patients who had had a prior null response received Faldaprevir 240mg once daily, in the form of 2 soft gelatin capsules administered orally, combined with PegIFN/RBV, administered by injection, for 12 weeks, followed by placebo once daily combined with PegIFN/RBV for 12 weeks. Followed by PegIFN/RBV alone for 24 weeks.
- Null:Faldaprevir 24 Weeks: Patients who had had a prior null response received Faldaprevir 240mg once daily, in the form of 2 soft gelatin capsules administered orally, combined with PegIFN/RBV, administered by injection, for 24 weeks. Followed by PegIFN/RBV alone for 24 weeks.
Period: Overall Study
Arm/Group | Relapser:Placebo | Relapser:Faldaprevir 12 Weeks | Relapser:Faldaprevir 24 Weeks | Partial:Placebo | Partial:Faldaprevir 12 Weeks | Partial:Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks
Started | 49 | 99 | 103 | 29 | 57 | 55 | 146 | 140
Completed | 18 | 86 | 87 | 10 | 46 | 42 | 81 | 85
Not Completed | 31 | 13 | 16 | 19 | 11 | 13 | 65 | 55
Not completed — Adverse Event | 0 | 6 | 9 | 0 | 4 | 8 | 12 | 7
Not completed — Lack of Efficacy | 26 | 3 | 4 | 19 | 7 | 4 | 49 | 44
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 4 | 2 | 0 | 0 | 1 | 1 | 3
Not completed — Other reason not defined above | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Not treated | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS)
Groups:
- Relapser:Faldaprevir 12 Weeks: Patients who had had a prior relapse, received Faldaprevir 240mg once daily, in the form of 2 soft gelatin capsules administered orally, combined with PegIFN/RBV, administered by injection, for 12 weeks, followed by placebo once daily combined with PegIFN/RBV for 12 weeks. At week 24, if the patients did not achieve early treatment success (ETS) the patients received an additional 24 weeks of PegIFN/RBV alone.
- Total: Total of all reporting groups
Arm/Group | Relapser:Placebo | Relapser:Faldaprevir 12 Weeks | Relapser:Faldaprevir 24 Weeks | Partial:Placebo | Partial:Faldaprevir 12 Weeks | Partial:Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks | Total
Number analyzed (Participants) | 49 | 99 | 103 | 29 | 57 | 55 | 145 | 140 | 677
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (8.29) | 53.5 (8.57) | 53.7 (8.14) | 55.7 (7.50) | 52.7 (7.90) | 52.0 (10.32) | 53.2 (8.76) | 53.6 (8.13) | 53.4 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 44 | 43 | 10 | 20 | 20 | 54 | 63 | 274
  Male | 29 | 55 | 60 | 19 | 37 | 35 | 91 | 77 | 403

OUTCOME MEASURES:

1. Secondary Outcome: Virological Response After 24 Weeks of Treatment Discontinuation (SVR24)
Description: Percentage of participants with virological response after 24 weeks of treatment discontinuation (SVR24) defined as plasma Hepatitis C virus Ribonucleic acid (HCV RNA) level <25 IU/mL (undetected) 24 weeks after the originally planned treatment duration.
Time Frame: 24 weeks post treatment, up to 72 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Relapser & Partial: Placebo: Patients who had had a prior relapse or prior partial response, received 2 soft gelatin capsules identical to those containing Faldaprevir once daily (orally) and PegIFN/RBV administered by injection, for 24 weeks, followed by PegIFN/RBV for 24 weeks.
- Relapser & Partial: Faldaprevir 12 Weeks: Patients who had had a prior relapse or prior partial response, received Faldaprevir 240mg once daily, in the form of 2 soft gelatin capsules administered orally, combined with PegIFN/RBV, administered by injection, for 12 weeks, followed by placebo once daily combined with PegIFN/RBV for 12 weeks. Followed by PegIFN/RBV alone for 24 weeks (for the partial relapsers the last 24 weeks was only if the patient did not achieve early treatment success (ETS)).
- Relapser & Partial: Faldaprevir 24 Weeks: Patients who had had a prior relapse or prior partial response, received Faldaprevir 240mg once daily, in the form of 2 soft gelatin capsules administered orally, combined with PegIFN/RBV, administered by injection, for 24 weeks. Followed by PegIFN/RBV alone for 24 weeks (for the partial relapsers the last 24 weeks was only if the patient did not achieve early treatment success (ETS)).
Arm/Group | Relapser & Partial: Placebo | Relapser & Partial: Faldaprevir 12 Weeks | Relapser & Partial: Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks
Number analyzed (Participants) | 78 | 156 | 158 | 145 | 140
percentage of participants | 10.3 [3.5 to 17.0] | 63.5 [55.9 to 71.0] | 59.5 [51.8 to 67.1] | 33.8 [26.1 to 41.5] | 32.9 [25.1 to 40.6]
Statistical Analysis 1: Comparison: Relapser & Partial: Placebo vs Relapser & Partial: Faldaprevir 12 Weeks; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Adjusted for genotype and previous response to treatment; Adjusted percent difference = 52.8, 95% CI 2-sided [42.4 to 63.2]
Statistical Analysis 2: Comparison: Relapser & Partial: Placebo vs Relapser & Partial: Faldaprevir 24 Weeks; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Adjusted for genotype and previous response to treatment; Adjusted percent difference = 48.5, 95% CI 2-sided [38.2 to 58.9]
Statistical Analysis 3: Comparison: Relapser & Partial: Faldaprevir 12 Weeks vs Relapser & Partial: Faldaprevir 24 Weeks; Test type: Superiority or Other; Adjusted percent difference = 4.4, 95% CI 2-sided [-6.0 to 14.9]
Statistical Analysis 4: Comparison: Null:Faldaprevir 12 Weeks vs Null:Faldaprevir 24 Weeks; Test type: Superiority or Other; Adjusted percent difference = -0.1, 95% CI 2-sided [-10.9 to 10.7]
Statistical Analysis 5: Comparison: Null:Faldaprevir 12 Weeks; Comparison is based on the Null:Faldaprevir 12 weeks vs historical rate of 20%; Test type: Superiority or Other; p < 0.0001, Normal approximation
Statistical Analysis 6: Comparison: Null:Faldaprevir 24 Weeks; Comparison is based on the Null:Faldaprevir 24 weeks vs historical rate of 20%; Test type: Superiority or Other; p = 0.0001, Normal approximation

2. Secondary Outcome: Early Treatment Success (ETS)
Description: Percentage of participants with early Treatment Success (ETS) defined as a plasma HCV RNA level <25 IU/mL (undetected or detected) at Week 4 and <25 IU/mL (undetected) at Week 8.
Time Frame: Week 4 and Week 8
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Relapser:Placebo | Relapser:Faldaprevir 12 Weeks | Relapser:Faldaprevir 24 Weeks | Partial:Placebo | Partial:Faldaprevir 12 Weeks | Partial:Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks
Number analyzed (Participants) | 49 | 99 | 103 | 29 | 57 | 55 | 145 | 140
percentage of participants | 4.1 | 85.9 | 87.4 | 3.4 | 66.7 | 76.4 | 58.6 | 51.4

3. Primary Outcome: Sustained Virological Response 12 Weeks Post Treatment (SVR12)
Description: Percentage of participants with sustained virological response (SVR12) 12 weeks post treatment defined as plasma Hepatitis C virus Ribonucleic acid (HCV RNA) level <25 IU/mL (undetected) 12 weeks after the originally planned treatment duration.
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relapser & Partial: Placebo | Relapser & Partial: Faldaprevir 12 Weeks | Relapser & Partial: Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks
Number analyzed (Participants) | 78 | 156 | 158 | 145 | 140
percentage of participants | 10.3 [3.5 to 17.0] | 65.4 [57.9 to 72.9] | 61.4 [53.8 to 69.0] | 33.8 [26.1 to 41.5] | 32.9 [25.1 to 40.6]
Statistical Analysis 1: Comparison: Relapser & Partial: Placebo vs Relapser & Partial: Faldaprevir 12 Weeks; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Adjusted for genotype and previous response to treatment; Adjusted percent difference = 54.7, 95% CI 2-sided [44.4 to 65.0]
Statistical Analysis 2: Comparison: Relapser & Partial: Placebo vs Relapser & Partial: Faldaprevir 24 Weeks; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Adjusted for genotype and previous response to treatment; Adjusted percent difference = 50.4, 95% CI 2-sided [40.1 to 60.8]
Statistical Analysis 3: Comparison: Relapser & Partial: Faldaprevir 12 Weeks vs Relapser & Partial: Faldaprevir 24 Weeks; Test type: Superiority or Other; Adjusted percent difference = 4.5, 95% CI 2-sided [-5.8 to 14.9]
Statistical Analysis 4: Comparison: Null:Faldaprevir 12 Weeks vs Null:Faldaprevir 24 Weeks; Test type: Superiority or Other; Adjusted percent difference = -0.1, 95% CI 2-sided [-10.9 to 10.7]
Statistical Analysis 5: Comparison: Null:Faldaprevir 12 Weeks; Comparison is based on the Null:Faldaprevir 12 weeks vs historical rate of 20%; Test type: Superiority or Other; p < 0.0001, Normal approximation
Statistical Analysis 6: Comparison: Null:Faldaprevir 24 Weeks; Comparison is based on the Null:Faldaprevir 24 weeks vs historical rate of 20%; Test type: Superiority or Other; p = 0.0001, Normal approximation

4. Secondary Outcome: ALT Normalisation: ALT in Normal Range at End of Treatment, When SVR12=NO
Description: The number of participants with alanine aminotransferase (ALT) in normal range at the end of treatment (EoT) when patients do not have sustained virological response 12 weeks post treatment. BL=baseline
Time Frame: End of treatment, up to 48 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Relapser:Placebo | Relapser:Faldaprevir 12 Weeks | Relapser:Faldaprevir 24 Weeks | Partial:Placebo | Partial:Faldaprevir 12 Weeks | Partial:Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks
Number analyzed (Participants) | 49 | 99 | 103 | 29 | 57 | 55 | 145 | 140
participants
  SVR12=NO | 42 | 30 | 31 | 28 | 24 | 30 | 96 | 94
  BL normal to EoT normal | 9 | 9 | 6 | 3 | 4 | 4 | 15 | 14
  BL elevated to EoT normal | 15 | 10 | 14 | 9 | 14 | 6 | 34 | 38
  No EoT data available for ALT | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0

5. Secondary Outcome: ALT Normalisation: ALT in Normal Range at End of Treatment, When SVR12=YES
Description: The number of participants with alanine aminotransferase (ALT) in normal range at the end of treatment when patients have sustained virological response 12 weeks post treatment. BL=baseline
Time Frame: End of treatment, up to 48 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Relapser:Placebo | Relapser:Faldaprevir 12 Weeks | Relapser:Faldaprevir 24 Weeks | Partial:Placebo | Partial:Faldaprevir 12 Weeks | Partial:Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks
Number analyzed (Participants) | 49 | 99 | 103 | 29 | 57 | 55 | 145 | 140
participants
  SVR12=YES | 7 | 69 | 72 | 1 | 33 | 25 | 49 | 46
  BL normal to EoT normal | 3 | 30 | 30 | 0 | 10 | 8 | 12 | 9
  BL elevated to EoT normal | 4 | 29 | 26 | 1 | 14 | 8 | 23 | 27

6. Secondary Outcome: AST Normalisation: AST in Normal Range at End of Treatment, When SVR12=NO
Description: The number of participants with aspartate aminotransferase (AST) in normal range at the end of treatment when patients do not have sustained virological response 12 weeks post treatment. BL=baseline
Time Frame: End of treatment, up to 48 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Relapser:Placebo | Relapser:Faldaprevir 12 Weeks | Relapser:Faldaprevir 24 Weeks | Partial:Placebo | Partial:Faldaprevir 12 Weeks | Partial:Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks
Number analyzed (Participants) | 49 | 99 | 103 | 29 | 57 | 55 | 145 | 140
participants
  SVR12=NO | 42 | 30 | 31 | 28 | 24 | 30 | 96 | 94
  BL normal to EoT normal | 19 | 16 | 12 | 4 | 3 | 5 | 18 | 21
  BL elevated to EoT normal | 5 | 5 | 9 | 9 | 14 | 6 | 24 | 28

7. Secondary Outcome: AST Normalisation: AST in Normal Range at End of Treatment, When SVR12=YES
Description: The number of participants with aspartate aminotransferase (AST) in normal range at the end of treatment (EoT) when patients have sustained virological response 12 weeks post treatment. BL=baseline
Time Frame: End of treatment, up to 48 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Relapser:Placebo | Relapser:Faldaprevir 12 Weeks | Relapser:Faldaprevir 24 Weeks | Partial:Placebo | Partial:Faldaprevir 12 Weeks | Partial:Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks
Number analyzed (Participants) | 49 | 99 | 103 | 29 | 57 | 55 | 145 | 140
participants
  SVR12=YES | 7 | 69 | 72 | 1 | 33 | 25 | 49 | 46
  BL normal to EoT normal | 2 | 35 | 39 | 0 | 13 | 10 | 15 | 16
  BL elevated to EoT normal | 4 | 24 | 22 | 1 | 10 | 9 | 21 | 20
  No EoT data available for AST | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0

8. Secondary Outcome: ALT Normalisation: ALT in Normal Range 12 Weeks Post Treatment, When SVR12=NO
Description: The number of participants with alanine aminotransferase (ALT) in normal range post treatment when patients do not have sustained virological response 12 weeks post treatment. BL=baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Relapser:Placebo | Relapser:Faldaprevir 12 Weeks | Relapser:Faldaprevir 24 Weeks | Partial:Placebo | Partial:Faldaprevir 12 Weeks | Partial:Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks
Number analyzed (Participants) | 49 | 99 | 103 | 29 | 57 | 55 | 145 | 140
participants
  SVR12=NO | 42 | 30 | 31 | 28 | 24 | 30 | 96 | 94
  BL normal to SVR12 normal | 0 | 9 | 6 | 0 | 2 | 4 | 11 | 6
  BL elevated to SVR12 normal | 1 | 6 | 6 | 0 | 4 | 3 | 7 | 9
  No ALT data available at SVR12 visit | 33 | 7 | 3 | 23 | 6 | 5 | 27 | 30

9. Secondary Outcome: ALT Normalisation: ALT in Normal Range 12 Weeks Post Treatment, SVR12=YES
Description: The number of participants with alanine aminotransferase (ALT) in normal range post treatment when patients have sustained virological response 12 weeks post treatment. BL=baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Relapser:Placebo | Relapser:Faldaprevir 12 Weeks | Relapser:Faldaprevir 24 Weeks | Partial:Placebo | Partial:Faldaprevir 12 Weeks | Partial:Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks
Number analyzed (Participants) | 49 | 99 | 103 | 29 | 57 | 55 | 145 | 140
participants
  SVR12=YES | 7 | 69 | 72 | 1 | 33 | 25 | 49 | 46
  BL normal to SVR12 normal | 3 | 31 | 31 | 0 | 13 | 10 | 13 | 10
  BL elevated to SVR12 normal | 3 | 35 | 38 | 1 | 20 | 11 | 32 | 35
  No ALT data available at SVR12 visit | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0

10. Secondary Outcome: AST Normalisation: AST in Normal Range 12 Weeks Post Treatment, When SVR12=NO
Description: The number of participants with aspartate aminotransferase (AST) in normal range post treatment when patients do not have sustained virological response 12 weeks post treatment. BL=baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Relapser:Placebo | Relapser:Faldaprevir 12 Weeks | Relapser:Faldaprevir 24 Weeks | Partial:Placebo | Partial:Faldaprevir 12 Weeks | Partial:Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks
Number analyzed (Participants) | 49 | 99 | 103 | 29 | 57 | 55 | 145 | 140
participants
  SVR12=NO | 42 | 30 | 31 | 28 | 24 | 30 | 96 | 94
  BL normal to SVR12 normal | 0 | 14 | 10 | 0 | 3 | 3 | 13 | 14
  BL elevated to SVR12 normal | 2 | 2 | 6 | 0 | 6 | 3 | 6 | 3
  No AST data available at SVR12 visit | 33 | 7 | 3 | 23 | 6 | 6 | 27 | 30

11. Secondary Outcome: AST Normalisation: AST in Normal Range 12 Weeks Post Treatment, SVR12=YES
Description: The number of participants with aspartate aminotransferase (AST) in normal range post treatment when patients have sustained virological response 12 weeks post treatment. BL=baseline
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: FAS
Measure: Number; unit: participants
Arm/Group | Relapser:Placebo | Relapser:Faldaprevir 12 Weeks | Relapser:Faldaprevir 24 Weeks | Partial:Placebo | Partial:Faldaprevir 12 Weeks | Partial:Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks
Number analyzed (Participants) | 49 | 99 | 103 | 29 | 57 | 55 | 145 | 140
participants
  SVR12=YES | 7 | 69 | 72 | 1 | 33 | 25 | 49 | 46
  BL normal to SVR12 normal | 2 | 36 | 41 | 0 | 16 | 13 | 16 | 17
  BL elevated to SVR12 normal | 4 | 29 | 28 | 1 | 16 | 8 | 28 | 25
  No AST data available at SVR12 visit | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: During the course of the study (48 weeks)
Arm/Group | Relapser & Partial: Placebo | Relapser & Partial: Faldaprevir 12 Weeks | Relapser & Partial: Faldaprevir 24 Weeks | Null:Faldaprevir 12 Weeks | Null:Faldaprevir 24 Weeks
Serious Adverse Events (participants affected / at risk) | 1/78 | 14/156 | 13/158 | 16/145 | 11/140
Other Adverse Events (participants affected / at risk) | 74/78 | 148/156 | 156/158 | 142/145 | 139/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relapser & Partial: Placebo (N=78) | Relapser & Partial: Faldaprevir 12 Weeks (N=156) | Relapser & Partial: Faldaprevir 24 Weeks (N=158) | Null:Faldaprevir 12 Weeks (N=145) | Null:Faldaprevir 24 Weeks (N=140)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Keratosis follicular (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Oral lichen planus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Salivary gland calculus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 3 | 1 | 3 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 0
International normalised ratio abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Coma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Psychiatric decompensation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Traumatic haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relapser & Partial: Placebo (N=78) | Relapser & Partial: Faldaprevir 12 Weeks (N=156) | Relapser & Partial: Faldaprevir 24 Weeks (N=158) | Null:Faldaprevir 12 Weeks (N=145) | Null:Faldaprevir 24 Weeks (N=140)
Anaemia (Blood and lymphatic system disorders) | 8 | 30 | 27 | 22 | 19
Neutropenia (Blood and lymphatic system disorders) | 12 | 18 | 18 | 16 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 4 | 6 | 13 | 3
Vertigo (Ear and labyrinth disorders) | 3 | 4 | 4 | 6 | 9
Dry eye (Eye disorders) | 5 | 6 | 7 | 4 | 5
Ocular icterus (Eye disorders) | 0 | 8 | 6 | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 8 | 14 | 7 | 13
Abdominal pain upper (Gastrointestinal disorders) | 4 | 16 | 15 | 11 | 15
Constipation (Gastrointestinal disorders) | 3 | 14 | 8 | 7 | 7
Diarrhoea (Gastrointestinal disorders) | 10 | 45 | 59 | 39 | 47
Dyspepsia (Gastrointestinal disorders) | 6 | 13 | 13 | 12 | 9
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 3 | 0 | 3 | 6
Nausea (Gastrointestinal disorders) | 18 | 78 | 88 | 77 | 75
Vomiting (Gastrointestinal disorders) | 5 | 41 | 47 | 46 | 37
Asthenia (General disorders) | 21 | 28 | 28 | 24 | 28
Chills (General disorders) | 5 | 9 | 14 | 1 | 8
Fatigue (General disorders) | 16 | 53 | 59 | 45 | 47
Influenza like illness (General disorders) | 15 | 28 | 29 | 27 | 23
Injection site erythema (General disorders) | 4 | 1 | 3 | 4 | 4
Malaise (General disorders) | 4 | 5 | 10 | 4 | 11
Pain (General disorders) | 4 | 5 | 7 | 4 | 4
Pyrexia (General disorders) | 14 | 24 | 25 | 26 | 38
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 11 | 11 | 10 | 9
Jaundice (Hepatobiliary disorders) | 1 | 29 | 27 | 16 | 16
Influenza (Infections and infestations) | 4 | 4 | 6 | 4 | 1
Nasopharyngitis (Infections and infestations) | 7 | 14 | 13 | 6 | 10
Haemoglobin decreased (Investigations) | 2 | 6 | 4 | 9 | 10
Weight decreased (Investigations) | 3 | 7 | 2 | 8 | 8
Decreased appetite (Metabolism and nutrition disorders) | 10 | 33 | 32 | 27 | 36
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 14 | 21 | 10 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 14 | 12 | 5 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 7 | 8 | 4 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 20 | 19 | 15 | 18
Disturbance in attention (Nervous system disorders) | 1 | 4 | 9 | 2 | 4
Dizziness (Nervous system disorders) | 6 | 12 | 11 | 9 | 5
Dysgeusia (Nervous system disorders) | 4 | 8 | 12 | 7 | 12
Headache (Nervous system disorders) | 22 | 39 | 46 | 52 | 45
Anxiety (Psychiatric disorders) | 3 | 9 | 12 | 5 | 11
Depression (Psychiatric disorders) | 10 | 11 | 12 | 14 | 15
Insomnia (Psychiatric disorders) | 13 | 36 | 35 | 18 | 29
Sleep disorder (Psychiatric disorders) | 3 | 4 | 5 | 8 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 25 | 27 | 23 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 16 | 16 | 8 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3 | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 16 | 16 | 8 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 29 | 29 | 19 | 31
Erythema (Skin and subcutaneous tissue disorders) | 4 | 8 | 9 | 11 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 23 | 54 | 61 | 47 | 63
Rash (Skin and subcutaneous tissue disorders) | 16 | 37 | 44 | 38 | 41
Irritability (Psychiatric disorders) | 11 | 10 | 16 | 10 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.